CLINICAL TRIAL: NCT05143372
Title: The Effect of Various Modes of Vibroacoustic Therapy on the Course of Coronavirus Infection Complicated by Acute Respiratory Failure.
Brief Title: Influence of Vibroacoustic Therapy Modes on the Course of Coronavirus Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astana Medical University (Other)
Responsible Party: Principal Investigator, Aidos Konkayev, professor, Astana Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: СТЛ-000215
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Acute Respiratory Failure; Vibration; Exposure
Keywords: Acute Respiratory Failure; Vibration; Exposure; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SaO2 (oxygen status) (Active Comparator): Measurment 4 times per day, ABA (acid-bases analyses)
  Interventions: Device: Vibrolung
- PaO2/FiO2 (respiratory index) (Active Comparator): Measurment 4 times per day, ABA (acid-bases analyses)
  Interventions: Device: Vibrolung

INTERVENTIONS:
Device: Vibrolung — Vibroacoustic respiratory therapy

SUMMARY:
Assessment of the dynamics of changes in physical, instrumental and laboratory parameters in patients with identified coronavirus infection complicated by acute respiratory failure included in the study in accordance with the inclusion criteria, and comparison of the results with the control group, study of the effect of modes when using vibroacoustic lung therapy.

ELIGIBILITY:
Inclusion Criteria:

* adults
* P/F less 300 torr
* COVID-19 Virus Infection

Exclusion Criteria:

* children
* acute stroke
* acute coronary syndrome
* DVT
* implanted pacemaker
* rib fracture
* infection on chest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change of time spent on ventilation | 1-2 days
  Changing of the time spent by patients on mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (3):
- Kazakhstan (3):
  - NATIONAL CENTER Scientific Center of Traumatology and Orthopedics named after Academician Batpenov N.D., Astana
  - Multidisciplinary city hospital No. 3 of Nursultan, Astana
  - Multidisciplinary Infectious Diseases Hospital of Nursultan, Astana

REFERENCES:
- [Derived] Konkayev A, Bekniyazova A. Vibroacoustic therapy in the treatment of patients with COVID-19 complicated by respiratory failure: a pilot randomized controlled trial. Front Med (Lausanne). 2023 Dec 14;10:1225384. doi: 10.3389/fmed.2023.1225384. eCollection 2023. PMID 38155668